| 'Development of isthmocele symptom severity and quality of life scale' |
|------------------------------------------------------------------------|
| NCT Number: |
| 01.01.2023 |

Isthmocele, also known as a cesarean scar defect, is the disruption of the integrity of the myometrium in the cesarean section incision and the indentation of the opening in the myometrium towards the visceral peritoneum. Residual menstrual blood accumulating in the isthmocele sac can cause chronic endometritis, abnormal uterine bleeding, infertility, and chronic pelvic pain. There is currently no quality of life scale that assesses isthmocele symptoms. A scale is needed to determine the effect on the patient's quality of life after the surgeries are performed. This study it is aimed to develop a scale that evaluates the severity of isthmocele symptoms and the impact on quality of life due to isthmocele. Patients with isthmocele symptoms three months after cesarean delivery will be included in the study. The study will not include findings that may be confused with isthmocele symptoms, such as uterine fibroids and endometrial polyps. Patients with acute vaginitis and pelvic inflammatory disease will not be included in the study. This study will be conducted on women diagnosed with symptomatic isthmocele after cesarean section. Researchers will prepare scale questions, and the survey questions will be developed after obtaining an expert opinion from 20 experts to be evaluated by psychiatry, obstetrics, and public health experts. The patient will fill out the questionnaire form with the diagnosis of isthmocele. Oral and written consent will be obtained from the patients. In the literature review, there is currently no quality of life scale for isthmocele symptoms. A scale is needed to detect changes in patients' quality of life after surgery due to isthmocele. This study aimed to create a questionnaire to evaluate the severity of isthmocele symptoms and the effect of isthmocele on quality of life.